CLINICAL TRIAL: NCT01427582
Title: YONDELIS(Trabectedin) Single Patient Compassionate Use / Expanded Access in Soft Tissue Sarcoma
Brief Title: YONDELIS (Trabectedin) Single Patient Compassionate Use / Expanded Access
Status: No longer available | Type: Expanded Access
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Other Study IDs: 05- EAP- STS
Record Dates: First submitted 2011-08-30; First posted 2011-09-01 (Estimated); Last update posted 2011-09-01 (Estimated); Status verified 2011-08

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Trabectedin

INTERVENTIONS:
Drug: Trabectedin — Trabectedin i.v. formulation at a dose of 1.5 mg/m2 i.v. over 24 hours on Day 1 every 21 days
  Other Names: YONDELIS

SUMMARY:
The YONDELIS (trabectedin) Single Patient Compassionate Use /Expanded Access program provides patients with advanced soft tissue sarcoma, who do not qualify for ongoing clinical trials with YONDELIS (trabectedin), access to this investigational treatment.

DETAILED DESCRIPTION:
The single patient treatment instructions for use are intended for a single patient with advanced soft tissue sarcoma. The patient will be treated with YONDELIS® (trabectedin) i.v. formulation at a dose of 1.5 mg/m2 i.v. over 24 hours on Day 1 every 21 days, provided that he/she fulfills all eligibility criteria.

The patient may continue to receive therapy until there is evidence of disease progression or unacceptable toxicity. Safety will be evaluated and serious adverse events will be reported. Disease assessments will occur according to institutional practice.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. 18 years-of-age or older.
3. Unresectable, advanced or metastatic, histologically proven soft tissue sarcoma.
4. Recovery from toxic effects of prior therapies to NCI CTC Grade 1 or better.
5. Hematologic variables:

   * Hemoglobin ≥9 g/dL
   * ANC ≥1,500/μL
   * Platelet count ≥100,000/μL
6. Serum creatinine ≤ upper limit of normal (ULN)
7. Hepatic function variables:

   * Total bilirubin ≤ ULN
   * Total alkaline phosphatase ≤ ULN, or if > ULN, then alkaline phosphatase liver fraction or 5'-nucleotidase must be ≤ ULN.
   * AST (serum aspartate transaminase [SGOT]) and ALT (serum alanine transaminase [SGPT]) must be ≤ 2.5xULN
   * Albumin ≥2.5 g/dL

Exclusion Criteria:

1. Pregnant or breast-feeding women, or patients (male or female) not employing adequate contraception. Acceptable means of birth control include IUD, oral contraceptive, subdermal implant, and a condom with a contraceptive sponge or suppository.
2. Less than 4 weeks from last dose of systemic cytotoxic therapy, radiation therapy, or therapy with any investigational agent
3. Active viral hepatitis or chronic liver disease
4. Unstable cardiac condition, including congestive heart failure or angina pectoris, myocardial infarction within 1 year before enrollment, uncontrolled arterial hypertension or arrhythmias
5. Active infection

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: John C. Bagwell, MD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Southwestern, Dallas, Texas, United States